CLINICAL TRIAL: NCT06629727
Title: The Effect Of Virtual Realty Glasses On Pain And Anxiety During The Kidney Stone Lithotripsy Procedure
Brief Title: The Effect Of Virtual Reality Glasses On Pain And Anxiety During The Kidney Stone Lithotripsy Procedure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Aysegul Gunes, Health Science Faculty Vice - Dean (PhD. RN.), University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Istanbul Beykent University
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Pain Management; Extracorporeal Shock Wave Lithotripsy; Virtual Reality
Keywords: extracorporeal shock wave lithotripsy; pain; Virtual reality; Anxiety
MeSH Terms: conditions — Agnosia; Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Use of VR glasses during the procedure
  Interventions: Other: VR Group
- Control Group (Active Comparator): Standart care group
  Interventions: Other: Control group

INTERVENTIONS:
Other: VR Group — the experimental group was shown a video through VRG during the lithotripsy procedure.
  Arms: VR group
Other: Control group — Patients received standard care during the procedure
  Arms: Control Group

SUMMARY:
To determine the pain and anxiety levels of patients using virtual reality glasses during the extracorporeal shock wave lithotripsy procedure.

DETAILED DESCRIPTION:
This randomized clinical trial included 60 patients with lithotripsy procedure. The research group of 60 people was divided into two groups, 30 in the experimental group and 30 in the control group. While the standard stone crushing process was applied to the control group, the experimental group was watched with virtual reality glasses during the procedure. The State-Trait Anxiety Inventory and the Numerical Rating Scale, which was used to measure the level of pain and anxiety level.

ELIGIBILITY:
Inclusion criteria

- Performing ESWL procedure

Exclusion criteria

* Presence of psychiatric disease
* Vision problem
* Hearing problem
* Drug and alcohol addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale | During ESWL procedure
  Pain level during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This was a masters thesis research, and the computer used to collect data at that time was damaged.
  Communication could not be established with the statistician who conducted the data analysis.

REFERENCES:
- [Result] Guitynavard F, Azadvari M, Gholamnejad M, et al. Decreasing discomfort during shock-wave lithotripsy using transcutaneous electrical nerve stimulation. Translational Research in Urology. 2022; 4(2): 71-76
- [Result] Lei M, Li G, Tang Y, Yuan J, Yang T, Gao Z. Efficacy of music therapy for pain control of extracorporeal shock wave lithotripsy: A meta-analysis of randomized controlled studies. Medicine (Baltimore). 2024 May 31;103(22):e38182. doi: 10.1097/MD.0000000000038182. PMID 39259054
- [Result] Ozsaker E, Diramali A. The effect of transcutaneous electrical nerve stimulation for pain relief during extracorporeal shock-wave lithotripsy procedure. Pain Manag Nurs. 2014 Mar;15(1):59-68. doi: 10.1016/j.pmn.2012.06.003. Epub 2012 Aug 18. PMID 24602425
- See also: The effect of transcutaneous electrical nerve stimulation for pain relief during extracorporeal shock-wave lithotripsy procedure. — https://doi.org/10.1016/j.pmn.2012.06.003
- See also: Impact of music on anxiety and pain control during extracorporeal shockwave lithotripsy: A protocol for systematic review and meta-analysis. — https://doi.org/10.1097/md.0000000000023684